CLINICAL TRIAL: NCT02004353
Title: Cochlear-Implanted Recipient Observational Study
Brief Title: Observation of Benefits for Patients Implanted With a Hearing Implant of the Company Cochlear
Acronym: IROS
Status: Terminated | Type: Observational
Why Stopped: Original study purpose accomplished
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL 5277
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2020-11

CONDITIONS: Hearing Loss
Keywords: Cochlear® Hearing Implants
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cochlear® Hearing Implants, hearing loss: Implanted Adolescents and Adults with permanent hearing loss
  Interventions: Device: Cochlear® Hearing Implants

INTERVENTIONS:
Device: Cochlear® Hearing Implants — Market approved hearing implants including: Nucleus Cochlear implants, Nucleus Auditory Brainstem Implants, Cochlear Baha implants, Cochlear Acoustic Implants

SUMMARY:
The purpose of this study is to collect patient related benefit data following treatment for permanent hearing loss with a hearing implant from the company Cochlear over a period of 2 years post treatment.

Assessment of benefits is based on standard questionnaires of hearing ability and quality of life in general.

DETAILED DESCRIPTION:
The clinical investigation is designed as a prospective repeated measures longitudinal study with intra-subject controls, using a selection of subjective evaluation tools to assess patient related benefits from hearing implant treatment of permanent hearing loss.

Clinically standard self-assessment scales, threshold measures and a general hearing history profile questionnaires for the clinician and implant recipient are made available for selection through an interface to a central electronic platform.

The registry is aimed at collection of data for patients who have already made the decision together with their implant centre clinician for an implant device from the company Cochlear.

Patients are approached for registry participation following implant by the caring clinician on a consecutive and voluntary basis and on condition of signing the patient informed consent.

Monitoring of data entry is included through automated reminders via e-platform and through inherent audit trail.

ELIGIBILITY:
Inclusion Criteria:

* Post-lingually deafened adults and adolescents who are newly implanted AND prior to first switch-on of their external device
* Unilateral, bilateral simultaneous recipients of any implant device(s) available with market approval from the company Cochlear®
* Children 10 years or older and in accordance with local regulations and product labelling
* Mentally capable to respond to self-administered assessment scales
* Willingness to participate and sign the Patient Informed Consent form

Exclusion Criteria:

* Individuals excluded from participation in a registry according to national or local regulations

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care routine clinical patients, with permanent hearing loss seeking implant treatment for hearing rehabilitation. Adolescent and Adult patients have limited or no benefit from conventional acoustic hearing aids.
Sampling Method: Non-Probability Sample
Enrollment: 1518 (Actual)
Dates: Start 2011-07; Primary Completion 2020-06-23 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Volckaerts, Study Director — Cochlear
Locations (77):
- Argentina (4):
  - Centro de Implantes Cocleares, Buenos Aires
  - Implantes Cocleares Equipo Multicentrico (ICEM), Buenos Aires
  - Centro de Investigaciones Otoaudiologicas (CIOA), Caba
  - Clinca Reina Fabiola, Córdoba
- Landesklinikum St. Pölten, Sankt Pölten, Austria
- University Hospital Leuven, Leuven, Belgium
- Hospital Edmundo Vasconcelos, São Paulo, Brazil
- Colombia (24):
  - Clinica Orlant, Antioquia
  - Te Oigo, Barranquilla
  - Clinica Rivas, Bogotá
  - Consultorio Gutierrez, Bogotá
  - Consultorio Navarro, Bogotá
  - Consultorio Ordonez, Bogotá
  - Consultorio Prieto, Bogotá
  - Consultório Plaza, Bogotá
  - DIAUDIO, Bogotá
  - Disaudio, Bogotá
  - Hospital de la Policia, Bogotá
  - Hospital San Jose Infantil, Bogotá
  - Hospital Universitario Clinica San Rafael, Bogotá
  - Instituto Nacional de Otologia Garcia Gomez, Bogotá
  - Mediglobal, Bogotá
  - Instituto para Niños Ciegos y Sordos, Cali
  - Consultório Velez, Cartagena
  - Consultório Mosquera, Ibagué
  - Consultorio Jaramillo, Manizales
  - Hospital Santa Sofia, Manizales
  - Clinica Sagrada Familia, Quindío
  - IPS San Rafael, Risaralda
  - Audiomedica, Santander
  - Consultorio Torres, Zipaquirá
- CHRU Lille, Lille, France
- Germany (10):
  - HNO Bad Aibling, Bad Aibling
  - Universitäts-Hals-Nasen-Ohren-Klinik Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinik für Hals-, Nasen- und Ohrenheilkunde, Freiburg im Breisgau
  - KMG Kliniken GmbH Güstrow, Güstrow
  - Medizinische Hochschule Hannover, Hanover
  - Helios München West, Münich
  - Eberhard-Karls-Universität Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - University of Wuerzburg, Würzburg
- University of Szeged, Szeged, Hungary
- Radboud University, Nijmegen, Netherlands
- Poland (11):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Uniwersytecki nr 2 w Bydgoszczy, Bydgoszcz
  - Wojewodzki Szpital Dzieciecy w Bydgoszczy, Bydgoszcz
  - World Hearing Center, Kajetany
  - Wojewodzki Szpital Zespolony w Koninie, Konin
  - Instytut Centrum Zdrowia Matki Polki w Lodzi, Lodz
  - Uniwersytecki Szpital Kliniczny nr 1 w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Wojewodzkie Centrum Medyczne w Opolu, Opole
  - Samodzielny Publiczny Szpital Kliniczny nr 2 w Poznaniu, Poznan
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Szczecinie, Szczecin
- Portugal (3):
  - CUF Infante Santo Hospital, Lisbon
  - Hospital Lusiadas Lisboa, Lisbon
  - Hospital CUF Porto, Porto
- UKC Maribor, Maribor, Slovenia
- South Africa (3):
  - Stellenbosch University, Cape Town
  - Durban Cochlear Implant Pogramme, Parklands Hospital, Durban
  - Johannesburg Cochlear Implant Center, Wits Donald Gordon Medical Centre, Johannesburg
- Spain (11):
  - Hospital de la Ribera, Alzira
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Donostia, Donostia / San Sebastian
  - Fundacion Jimenez Diaz, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinica Universitad de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario del Rio Hortega, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Karolinska Hospital Huddinge, Stockholm, Sweden
- Turkey (Türkiye) (3):
  - Osmangazi University Hospital, Eskişehir
  - Cerrahpasa University Hospital, Istanbul
  - Marmara University Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maes IH, Joore MA, Cima RF, Vlaeyen JW, Anteunis LJ. Assessment of health state in patients with tinnitus: a comparison of the EQ-5D and HUI mark III. Ear Hear. 2011 Jul-Aug;32(4):428-35. doi: 10.1097/AUD.0b013e3181fdf09f. PMID 21221004
- [Background] Noble W, Tyler R, Dunn C, Bhullar N. Unilateral and bilateral cochlear implants and the implant-plus-hearing-aid profile: comparing self-assessed and measured abilities. Int J Audiol. 2008 Aug;47(8):505-14. doi: 10.1080/14992020802070770. PMID 18608531
- [Derived] Mauch H, Kaur J, Irwin C, Wyss J. Design, implementation, and management of an international medical device registry. Trials. 2021 Nov 25;22(1):845. doi: 10.1186/s13063-021-05821-5. PMID 34823566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1518 participants were recruited in 77 centers from July 2011 to 31 July 2020
Groups:
- Cochlear® Hearing Implants: Nucleus Cochlear implants, Cochlear Baha implants, Cochlear Acoustic Implants
Period: Overall Study
Arm/Group | Cochlear® Hearing Implants
Started | 1518
Completed | 184
Not Completed | 1334
Not completed — Voluntary participation | 1334

BASELINE CHARACTERISTICS:
Population: Participants with baseline data recorded in the database.
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 1506
Age, Customized [Count of Participants; unit: Participants]
  <18 | 48
  18-34 | 351
  35-44 | 194
  45-54 | 268
  55-64 | 293
  >64 | 348
  Unknown | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 789
  Male | 717
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected.
Region of Enrollment [Number; unit: participants]
  Colombia | 396
  Argentina | 62
  Hungary | 47
  Portugal | 20
  Spain | 197
  Austria | 2
  Netherlands | 2
  Sweden | 3
  Turkey | 31
  Belgium | 7
  Poland | 193
  Brazil | 2
  South Africa | 200
  Slovenia | 16
  France | 36
  Germany | 292

OUTCOME MEASURES:

1. Primary Outcome: Change in Hearing Ability Assessed Via Speech Spatial Hearing Qualities Questionnaire
Description: A scale from 0 to 10 is used, where 0 represents "can not hear at all" and 10 "hear perfectly". The change from baseline to post-implant at 1 year is presented. A positive value indicates improved hearing, a negative value indicates impaired hearing.
Time Frame: Baseline (i.e. pre-implanted status, prior to 1st switch-on) and post-implant at 1 year
Population: For all devices with 50 or more participants with baseline data, analysis of the SSQ data was performed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 327
Score on a scale
  CI512 cochlear implant: number analyzed (Participants) | 133
  CI512 cochlear implant | 2.73 (0.148)
  CI522 cochlear implant: number analyzed (Participants) | 58
  CI522 cochlear implant | 2.1 (0.24)
  CI532 cochlear implant: number analyzed (Participants) | 60
  CI532 cochlear implant | 2.1 (0.27)
  Baha bone conduction hearing implant: number analyzed (Participants) | 76
  Baha bone conduction hearing implant | 2.2 (0.21)

2. Primary Outcome: Change in Hearing Ability Assessed Via Speech Spatial Hearing Qualities Questionnaire
Description: A scale from 0 to 10 is used, where 0 represents "can not hear at all" and 10 "hear perfectly". The change from baseline to post-implant at 2 years is presented. A positive value indicates improved hearing, a negative value indicates impaired hearing.
Time Frame: Baseline (i.e. pre-implanted status, prior to 1st switch-on) and post-implant at 2 years
Population: For all devices with 50 or more participants with baseline data, analysis of the SSQ data was performed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 160
Score on a scale
  CI512 cochlear implant: number analyzed (Participants) | 79
  CI512 cochlear implant | 2.95 (0.179)
  CI522 cochlear implant: number analyzed (Participants) | 32
  CI522 cochlear implant | 2.4 (0.31)
  CI532 cochlear implant: number analyzed (Participants) | 40
  CI532 cochlear implant | 2.5 (0.33)
  Baha bone conduction hearing implant: number analyzed (Participants) | 9
  Baha bone conduction hearing implant | 1.9 (0.65)

3. Primary Outcome: Change in Hearing Ability Assessed Via Speech Spatial Hearing Qualities Questionnaire
Description: A scale from 0 to 10 is used, where 0 represents "can not hear at all" and 10 "hear perfectly". The change from baseline to post-implant at 3 years is presented. A positive value indicates improved hearing, a negative value indicates impaired hearing.
Time Frame: Baseline (i.e. pre-implanted status, prior to 1st switch-on) and post-implant at 3 years
Population: For all devices with 50 or more participants with baseline data, analysis of the SSQ data was performed.There were too few Baha participants at years 3 to conduct a statistical analysis.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 69
Score on a scale
  CI512 cochlear implant: number analyzed (Participants) | 46
  CI512 cochlear implant | 2.74 (0.217)
  CI522 cochlear implant: number analyzed (Participants) | 17
  CI522 cochlear implant | 2.4 (0.39)
  CI532 cochlear implant: number analyzed (Participants) | 6
  CI532 cochlear implant | 2.6 (0.67)

4. Primary Outcome: Change in General Quality of Life Assessed Via Health Utility Index Mark III Questionnaire
Description: A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change from baseline to post-implant at 1 year is presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: Baseline (i.e. pre-implanted status, prior to 1st switch-on) and post-implant at 1 year
Population: For all devices with 50 or more participants with baseline data, analysis of the HUI3 data was performed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 327
Score on a scale
  CI512 cochlear implant: number analyzed (Participants) | 133
  CI512 cochlear implant | 0.166 (0.0212)
  CI522 cochlear implant: number analyzed (Participants) | 58
  CI522 cochlear implant | 0.22 (0.032)
  CI532 cochlear implant: number analyzed (Participants) | 60
  CI532 cochlear implant | 0.15 (0.034)
  Baha bone conduction hearing implant: number analyzed (Participants) | 76
  Baha bone conduction hearing implant | 0.12 (0.03)

5. Primary Outcome: Change in General Quality of Life Assessed Via Health Utility Index Mark III Questionnaire
Description: A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change from baseline to post-implant at 2 years is presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: Baseline (i.e. pre-implanted status, prior to 1st switch-on) and post-implant at 2 years
Population: For all devices with 50 or more participants with baseline data, analysis of the HUI3 data was performed.There were too few Baha participants at 2 years to conduct a statistical analysis.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 151
Score on a scale
  CI512 cochlear implant: number analyzed (Participants) | 79
  CI512 cochlear implant | 0.175 (0.0255)
  CI522 cochlear implant: number analyzed (Participants) | 32
  CI522 cochlear implant | 0.28 (0.04)
  CI532 cochlear implant: number analyzed (Participants) | 40
  CI532 cochlear implant | 0.15 (0.042)

6. Primary Outcome: Change in General Quality of Life Assessed Via Health Utility Index Mark III Questionnaire
Description: A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change from baseline to post-implant at 3 years is presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: Baseline (i.e. pre-implanted status, prior to 1st switch-on) and post-implant at 3 years
Population: For all devices with 50 or more participants with baseline data, analysis of the HUI3 data was performed.There were too few Baha participants at 3 years to conduct a statistical analysis.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 71
Score on a scale
  CI512 cochlear implant: number analyzed (Participants) | 48
  CI512 cochlear implant | 0.123 (0.0311)
  CI522 cochlear implant: number analyzed (Participants) | 17
  CI522 cochlear implant | 0.22 (0.051)
  CI532 cochlear implant: number analyzed (Participants) | 6
  CI532 cochlear implant | 0.27 (0.087)

7. Secondary Outcome: Unaided Hearing Thresholds
Description: Unaided hearing thresholds for bone and air conduction for the implanted and non-implanted ear to monitor clinically significant changes over time for frequencies between 500 Hz and 4000 Hz
Time Frame: Baseline (i.e. pre-implant status) assessed prior to 1st switch-on
Population: Results are for Baha participants. For the contra-lateral ear, data not received for all participants.
Measure: Mean (Standard Deviation); unit: Decibel
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 173
Decibel
  Air conduction-implanted ear | 71.7 (21.6)
  Bone conduction-implanted ear | 34.1 (24.4)
  Air conduction-contralateral year: number analyzed (Participants) | 168
  Air conduction-contralateral year | 36.7 (26.5)
  Bone conduction-contralateral ear: number analyzed (Participants) | 168
  Bone conduction-contralateral ear | 18.1 (15.7)

8. Secondary Outcome: Unaided Hearing Thresholds
Description: Unaided hearing thresholds for bone and air conduction for the implanted and non-implanted ear to monitor clinically significant changes over time for frequencies between 500 and 4000 Hz
Time Frame: post-implant at 1 year
Population: Results are for Baha participants. For the contra-lateral ear, data not received for all participants.
Measure: Mean (Standard Deviation); unit: Decibel
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 173
Decibel
  Air conduction-Implanted ear | 60.2 (24.2)
  Bone conduction-implanted ear | 29.4 (20.0)
  Air conduction- Contralateral ear: number analyzed (Participants) | 168
  Air conduction- Contralateral ear | 37.5 (24.5)
  Bone conduction-Contralateral ear: number analyzed (Participants) | 168
  Bone conduction-Contralateral ear | 18.1 (13.8)

9. Secondary Outcome: Unaided Hearing Thresholds
Description: Unaided hearing thresholds for bone and air conduction for the implanted and non-implanted ear to monitor clinically significant changes over time for frequencies between 125Hz and 8000 Hz
Time Frame: immediately post-implant
Population: Data not received due to voluntary participation of participants.
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 0

10. Secondary Outcome: Unaided Hearing Thresholds
Description: as for outcome 9
Time Frame: post-implant at 2 years
Population: Data not received due to voluntary participation of participants.
Arm/Group | Cochlear® Hearing Implants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Deaths, serious adverse events and non-serious adverse events were not assessed.
Arm/Group | Cochlear® Hearing Implants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-02-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT02004353/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT02004353/SAP_001.pdf